CLINICAL TRIAL: NCT06059196
Title: Adapting, Expanding, and Evaluating ARCHES (Addressing Reproductive Coercion in Health Settings) in Kenya
Brief Title: Adapting, Expanding and Evaluating ARCHES in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Population Council Kenya (Unknown); Kenya Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201922S
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Reproductive Coercion; Intimate Partner Violence
Keywords: Reproductive coercion; Intimate partner violence; Contraceptive Usage; Pregnancy Related; Quality of Care
MeSH Terms: conditions — Contraception Behavior | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial; stratified randomization based on facility type and urban/rural location.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Standard contraceptive counseling (Active Comparator): Standard contraceptive counseling, includes provider training on standard BCS+ counseling protocol and use of a companion mobile application to guide counseling
  Interventions: Behavioral: BCS+ (Balanced Counseling Strategy Plus)
- Intervention - Integrated contraceptive counseling (Experimental): Integrated contraceptive counseling, includes provider training on ARCHES integrated in BCS+ counseling protocol and use of a companion mobile application to guide counseling
  Interventions: Behavioral: ARCHES (Addressing Reproductive Coercion in Health Settings); Behavioral: BCS+ (Balanced Counseling Strategy Plus)

INTERVENTIONS:
Behavioral: ARCHES (Addressing Reproductive Coercion in Health Settings) — ARCHES (Addressing Reproductive Coercion in Health Settings) includes training existing contraceptive providers to (1) provide contraceptive clients with education on reproductive coercion and methods/ways to use contraceptive methods covertly if desired, (2) provide screening for reproductive coercion and intimate partner violence, (3) provide a referral to specialized services for those disclosing intimate partner violence, (4) and offer a palm-sized mini-booklet with educational information on reproductive coercion and intimate partner violence. A mobile application was developed to guide contraceptive providers through the counselling protocol.
  Arms: Intervention - Integrated contraceptive counseling
Behavioral: BCS+ (Balanced Counseling Strategy Plus) — BCS+ (Balanced Counseling Strategy Plus) is a contraceptive counseling protocol that contraceptive providers use to help clients identify suitable contraceptive methods based on their preferences and previous contraceptive experiences. The BCS+ also includes systematic screening for other health services such as HIV/STI, cervical cancer, and breast cancer. The BCS+ was adopted by the Kenya MOH as the standard contraceptive counseling protocol in the country.

SUMMARY:
Document evidence, via cluster randomized controlled trial, of the effectiveness of the ARCHES intervention, a brief, clinic-based counselling intervention demonstrated to reduce intimate partner violence and reproductive coercion and promote women's reproductive health, as scaled in government health facilities in Kenya, to (1) decrease unintended pregnancy, (2) increase family planning uptake and use/continuation, (3) decrease experiences of reproductive coercion and intimate partner violence of women and girls aged 15 to 49 years seeking family planning services, and, to (4) improve quality of care, (5) increase gender equitable attitudes, and, (6) increase self-efficacy to provide comprehensive family planning counseling among providers trained in ARCHES.

DETAILED DESCRIPTION:
Background: In Kenya, 17% of women have unmet need for family planning (FP) and the modern contraceptive prevalence rate (mCPR) has plateaued around 45%, contributing to poor reproductive health outcomes. This includes the nearly 50% of women in Kenya who report their last pregnancy as unintended, with those experiencing gender-based violence (GBV), particularly in the forms of intimate partner violence (IPV) and reproductive coercion (RC; behaviors that reduce women's ability to use contraception or otherwise prevent pregnancy), at significantly greater risk. Similar to other LMIC settings, both RC and IPV are highly prevalent in Kenya, particularly among women seeking FP and other reproductive health services (>1/3 of female FP clients). Since 2013, the World Health Organization (WHO) has strongly recommended that IPV and RC be addressed within reproductive health services and, in 2018, the Lancet Commission on Sexual and Reproductive Health and Rights found that RC and IPV were a significant contributor to unmet need for FP and unintended pregnancy, with greatest impacts among women and girls in LMICs. Within Kenya, the Ministry of Health (MOH) has made reduction of unintended pregnancy and gender-based violence (GBV), especially among adolescents, a primary objective. Despite this need and guidance, no clinic-based intervention models outside of the U.S. (apart from one, ARCHES) have demonstrated efficacy to improve FP uptake/use and reduce IPV or RC thereby reducing unintended pregnancy.

Intervention Description: ARCHES (Addressing Reproductive Coercion in Health Settings) is a brief, clinic-based intervention delivered by family planning providers aiming to: 1) Increase women's and girls' ability to use family planning in the face of reproductive coercion, facilitating women's voluntary family planning uptake and continued use without interference, 2) Provide a safe and supportive environment for IPV disclosure and subsequent referral to support services, and 3) Educate and support providers to improve quality of care related to family planning counseling, including addressing reproductive coercion and intimate partner violence.

Objective: The objective of this study is to generate evidence and learnings on scaling integrated family planning services (including family planning, reproductive coercion, and intimate partner violence) in public sector health facilities in Uasin Gishu County, Kenya via adaptation and implementation of ARCHES, in partnership with the Kenya MOH.

Methodology: A cluster randomized controlled trial paired with concurrent implementation science assessments will test effectiveness of the ARCHES model that has been adapted for scale by the Kenya MOH. Female family planning clients aged 15-49 years at selected sites will complete baseline surveys (immediately prior to receiving care), immediately post-visit exit surveys, and 6-month follow-up surveys. Family planning providers trained in ARCHES will complete pre-training, post-training, and 3-month follow-up surveys to assess changes in gender-equitable attitudes and self-efficacy to address issues of violence among their clients. Costs associated with the scale-up strategy will be tracked and utilized in combination with results of the effectiveness trial to assess total cost and cost-effectiveness of ARCHES.

ELIGIBILITY:
All eligibility criteria based on self-report.

Inclusion Criteria:

* Seeking family planning services at a selected study facility
* Aged 15-49 years old
* Female
* Able to provide informed consent
* Able to speak and understand English, Kiswahili, or Kalenjin
* Able to provide a safe phone number at which they can be recontacted for follow-up
* Not planning to move out of the area in the coming 6 months

Exclusion Criteria:

* Sterilized at baseline
* Pregnant at baseline

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — self-report biologically female
Enrollment: 3928 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Incident unintended pregnancy | 6-month follow-up
  Difference in self-reported unintended pregnancy in the past 6 months at the 6-month follow-up in intervention compared to control group (single time point analysis)

SECONDARY OUTCOMES:
Modern contraceptive use in the past 6 months | Baseline (at facility prior to receiving care) and 6-month follow-up
  Change in prevalence of self-reported modern contraceptive use in the past 6 months between baseline and 6-month follow-up in intervention compared to control group (difference-in differences)
Physical intimate partner violence in the past 6 months | Baseline (combined report at facility prior to receiving care and report at facility immediately after receiving care (post-visit); combined due to increased reporting post-visit) and 6-month follow-up
  Change in prevalence of self-reported physical intimate partner violence experience in the past 6 months between combined baseline/post-visit and 6-month follow-up in intervention compared to control group (difference-in differences)
Sexual intimate partner violence in the past 6 months | Baseline (combined report at facility prior to receiving care and report at facility immediately after receiving care (post-visit); combined due to increased reporting post-visit) and 6-month follow-up
  Change in prevalence of self-reported sexual intimate partner violence experience in the past 6 months between combined baseline/post-visit and 6-month follow-up in intervention compared to control group (difference-in differences)
Emotional intimate partner violence in the past 6 months | Baseline (combined report at facility prior to receiving care and report at facility immediately after receiving care (post-visit); combined due to increased reporting post-visit) and 6-month follow-up
  Change in prevalence of self-reported emotional intimate partner violence experience in the past 6 months between combined baseline/post-visit and 6-month follow-up in intervention compared to control group (difference-in differences)
Reproductive coercion from a male partner in the past 6 months | Baseline (combined report at facility prior to receiving care and report at facility immediately after receiving care (post-visit); combined due to increased reporting post-visit) and 6-month follow-up
  Change in prevalence of self-reported reproductive coercion experience in the past 6 months between combined baseline/post-visit and 6-month follow-up in intervention compared to control group (difference-in differences)
Incident pregnancy | 6-month follow-up
  Difference in self-reported pregnancy in the past 6 months at the 6-month follow-up in intervention compared to control group (single time point analysis)
Uptake of a modern contraceptive method | Post-visit (at facility immediately after receiving care)
  Difference in prevalence of self-reported modern contraceptive uptake post-visit in intervention compared to control group (single time point analysis)
Covert use of contraception in the past 6 months | Baseline (at facility prior to receiving care) and 6-month follow-up
  Change in prevalence of self-reported covert contraceptive use in the past 6 months between baseline and 6-month follow-up in intervention compared to control group (difference-in differences)
Contraceptive self-efficacy in the face of reproductive coercion | Baseline (at facility prior to receiving care), Post-visit (at facility immediately after receiving care), and 6-month follow-up
  Change in mean self-efficacy score (range: 3-9, higher=higher self-efficacy) between baseline, post-visit, and 6-month follow-up in intervention compared to control group (difference-in differences)
Awareness of intimate partner violence services | Baseline (at facility prior to receiving care), Post-visit (at facility immediately after receiving care), and 6-month follow-up
  Change in prevalence of awareness of intimate partner violence services between baseline, post-visit, and 6-month follow-up in intervention compared to control group (difference-in differences)
Self-efficacy to use intimate partner violence services | Baseline (at facility prior to receiving care), Post-visit (at facility immediately after receiving care), and 6-month follow-up
  Change in mean self-efficacy score (range: 1-3, higher=higher self-efficacy) between baseline, post-visit, and 6-month follow-up in intervention compared to control group (difference-in differences)
Use of intimate partner violence services | 6-month follow-up
  Difference in prevalence of use of intimate partner violence services in the past 6 months at the 6-month follow-up in intervention compared to control group (single time point analysis)
Attitudes accepting of reproductive coercion | Baseline (at facility prior to receiving care), Post-visit (at facility immediately after receiving care), and 6-month follow-up
  Change in mean attitude score (range: 6-12, higher=attitudes less accepting of reproductive coercion/improved attitudes) between baseline, post-visit, and 6-month follow-up in intervention compared to control group (difference-in differences)
Quality of family planning care | Post-visit (at facility immediately after receiving care)
  Difference in mean (range: 11-55, higher=higher quality) interpersonal quality of family planning scale post-visit in intervention compared to control group (single time point analysis)
Discontinuation of modern contraception | 6-month follow-up
  Difference in prevalence of modern contraceptive discontinuation in the past 6 months at the 6-month follow-up in intervention compared to control group (single time point analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Jay G Silverman, PhD, Principal Investigator — University of California, San Diego
Locations (24):
- Kenya (24):
  - Burnt Forest Sub-county Hospital, Burnt Forest
  - Kipkabus Health Centre, Burnt Forest
  - Chepkigen Health Centre, Cheptiret
  - Huruma District Hospital, Eldoret
  - Kapsoya Health Centre, Eldoret
  - Kapteldon Health Centre, Eldoret
  - Kapyemit Dispensary, Eldoret
  - Kipkenyo, Eldoret
  - Pioneer Health Centre, Eldoret
  - Railways, Eldoret
  - Uasin Gishu District Hospital, Eldoret
  - Kesses Health Centre, Kesses
  - Chembulet Health Centre, Kimumu
  - Chepkanga Health Centre, Kimumu
  - Merewet Dispensary, Kimumu
  - Moiben Health Centre, Moiben
  - Moi's Bridge Health Centre, Moi‘s Bridge
  - Chepkero Dispensary, Naiberi
  - Soy Health Centre, Soy
  - Sosiani Health Centre, Turbo
  - Turbo Sub-County Hospital, Turbo
  - Kabobo Health Centre, Ziwa
  - Kipsigak Health Centre, Ziwa
  - Ziwa Sub-County Hospital, Ziwa

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified participant data analysis sets to the Dyrad public data repository upon publication of findings
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication of findings
Access Criteria: Open access

REFERENCES:
- [Derived] Pearson E, Uysal J, Menzel J, Undie CC, Odwe G, Liambila W, Silverman JG. Evaluating a scalable ARCHES (Addressing Reproductive Coercion in Health Settings) model in government health facilities in Uasin Gishu county, Kenya: study protocol for a cluster-randomized controlled trial. Reprod Health. 2023 Oct 17;20(1):155. doi: 10.1186/s12978-023-01697-7. PMID 37848916